CLINICAL TRIAL: NCT06306053
Title: A New Digital Technology-based Treatment for Chronic Pain Combining Neuromodulation, Computerassisted Training and Telemonitoring
Brief Title: A New Treatment for Chronic Pain Combining Neuromodulation, Computer Assisted Training and Telemonitoring
Acronym: TechNoPain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Santi Paolo e Carlo (Other)
Collaborators: University of Milan (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Istituto Europeo di Oncologia (Other)
Responsible Party: Principal Investigator, Alberto Priori, Professor, ASST Santi Paolo e Carlo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/ST/217
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: neuromodulation; pain; telemonitoring; motor training; tDCS
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A Group (Experimental): Only tDCS treatment
  Interventions: Device: tDCS
- B Group (Active Comparator): Only Motor Training
  Interventions: Other: EuleriaLab
- C Group (Active Comparator): Both Treatment (tDCS+Motor Training)
  Interventions: Combination Product: tDCS+EuleriaLab

INTERVENTIONS:
Combination Product: tDCS+EuleriaLab — Home based: Non invasive Neuromodulation treatment + Motor Training
  Arms: C Group
Device: tDCS — Non invasive brain stimulation
  Arms: A Group
Other: EuleriaLab — Home Motor Training
  Arms: B Group

SUMMARY:
Chronic pain (CP) is a leading cause of medical disability, healthcare expenditure, and reduced psychological well-being. Given the limited mobility, travel burden, and cost, access to care can be problematic for patients suffering from this disease, driving the recent shift toward care through telehealth programs. Given the complex interrelationship of physical and psychosocial aspects related to chronic pain, in this project the investigators propose to validate and investigate the effectiveness of new integrated health interventions by combining the technique of transcranial direct current stimulation (tDCS), complementary therapies and telemonitoring. The investigators hypothesize that this novel combined approach will provide a more effective strategy to overcome the classic barriers of pharmacological treatments and access to healthcare due to lack of mobility. To do this, the investigators will rely on a previously developed integrated platform that enables effective delivery of non-pharmacological interventions and outcome assessment. Many patients do not benefit from pharmacological and invasive treatments, leading to the development of alternative therapeutic options such as non-invasive brain stimulation (e.g. tDCS) and complementary interventions to improve physical and psychological well-being. These complementary interventions reduced pain intensity and psychological distress by improving individuals' ability to manage and cope with their pain. However, due to the multiple co-occurring factors associated with chronic pain, a multidisciplinary and integrated treatment approach is challenging. Technology ecosystems can be a reliable tool to achieve such a diverse personalized approach and evaluate their results. In a previous project, the investigators developed PainRE-Life, a dynamic and integrated technology ecosystem to enable continuity of care for CP patients, including personalized applications, training tools and telemonitoring tools for outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic pain (Fibromyalgia, Headache, Oncological Pain)
* Age > 18;
* Cognitive and motor skills sufficient to support a rehabilitation process mediated by an electronic device on a signed declaration by the clinician; -Having completed and signed the informed consent form, after a detailed explanation of the task and the tools used in the study.

Exclusion Criteria:

* Have started new pharmacological treatments or have changed therapies that act on pain for less than a month;
* Have a brain stimulator, heart marrow stimulator or pumps for intrathecal drug delivery;
* Respiratory, cardiac, metabolic or other conditions incompatible with at least 30 minutes of light or moderate intensity exercise therapy;
* Aphasia, dementia, or psychiatric comorbidity interfering with communication or rehabilitation program compliance;
* Severe cognitive deficits;
* Blindness or severe vision problems which may interfere with the use of the tablet;
* Presence of cranial bone breaches;
* Recurrent seizures not being treated;
* Insufficient knowledge of the Italian language and/or inability to understand verbal and written instructions;
* Concomitant participation in another study or clinical trial involving rehabilitation therapy (recreational therapy, occupational therapy, physiotherapy) or administration of an investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best). The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
12-item Short Form Survey (SF12) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  Short Form Survey (SF-12) is a health-related quality of life assessment tool that measures patients' physical and mental health. The lowest possible value is 0 and the highest is 100. In general, the highest values indicate a better result and the lowest indicate a worse result.
Hospital Anxiety and Depression scale (HADS) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). 0-7 (Normal) 8-10 (Mild) 11-15 (Moderate) 16-21 (Severe)
Brief Pain Inventory (BPI) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  This self-administered questionnaire assesses pain severity and its impact on quality of life through 15 questions. The patients responded using a 10-point Likert scale, with higher scores indicating greater pain severity and greater interference with that aspect of life.
Pain Catastrophizing Scale (PCS) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  This self-administered questionnaire measures catastrophic thinking related to chronic pain. The patients rated how often they have 13 different thoughts and feelings while experiencing pain from 0 to 4. The total sum of the scores ranges between 0 and 52, with higher total scores indicating more catastrophic thinking.
Shared Decision-Making Questionnaire 9-Item (SDM-Q-9) | Baseline (Day 1), after 1 week of treatment (Day 5), at the end of the treatment (Day 19), one month follow up (month 1), 3 months follow up (month 3)
  The SDM-Q-9 instrument was developed to assess the patient subjective experience of SDM according to nine stages on the decision-making process. It describes the experience of SDM through nine items which are scored on a six-point Likert scale from 0 (completely disagree) to 5 (completely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Priori, PhD, Principal Investigator — ASST-Santi Paolo e Carlo Hospital
Locations (3):
- Italy (3):
  - ASST-Santi Paolo e Carlo Hospital, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Europeo di Oncologia, Milan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP